CLINICAL TRIAL: NCT02913898
Title: Dynamic Learning in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dynamic Learning in Depression
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2019-04

CONDITIONS: Depression
Keywords: learning
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IBLT (information bias learning task) (Experimental): Computerised task in which most information is provided by positive outcomes. Completed for 10 mins per day every day for 2 weeks.
  Interventions: Behavioral: IBLT
- IBLT control (Placebo Comparator): Computerised task in which information is provided by both positive and negative outcomes. Completed 10 mins per day every day for 2 weeks
  Interventions: Behavioral: IBLT control

INTERVENTIONS:
Behavioral: IBLT — Information bias learning task-- a computer based task in which positive information is more useful when learning how best to complete it
  Arms: IBLT (information bias learning task)
Behavioral: IBLT control — A control version of the IBLT task-- a computer based task in which both positive and negative information is useful when learning how to complete it
  Arms: IBLT control

SUMMARY:
This study will assess learning bias (the tendency to learn more from negative relative to positive outcomes) at baseline in 3 groups of participants (currently depressed, previously depressed and never depressed). It will then try to modify this bias using a simple computerised training task completed at home daily for 2 weeks. Outcome measures include symptoms of depression, cognitive measures (i.e. accuracy and reaction time during completion of tasks), pupillometry measures and salivary cortisol.

DETAILED DESCRIPTION:
Depressed patients tend to focus on negative, at the expense of positive, events. This bias of attention is thought to be one factor which causes some people to be at higher risk of developing depression. One reason depressed people might pay more attention to negative events is that they think those events are more useful to them when they learn about the future. In this study the investigators will compare the learning styles (i.e. whether participants focus more on negative or positive information when learning about the future), cognitive biases and salivary cortisol levels (the levels of the hormone cortisol can be measured in the saliva and is known to be raised in those at risk of depression) of currently depressed (N=40), previously depressed (N=40) and never depressed (N=40) participants. The study will then randomly assign participants to complete one of two version of a learning task daily over two weeks. One version of the task will be designed to encourage an optimistic learning style, whereas the other will encourage neither an optimistic nor pessimistic learning style. The study will then retest participants' learning styles, cognitive biases, salivary cortisol and mood (using questionnaire measures) after completion of the task and again after 1 month. Study activities for participants will be: Screening visit (1 hours), baseline test visit (2 hours), task completion at home (10 mins per day for 2 weeks), test visit 2 (2 hours, completed 2 weeks after baseline visit) and test visit 3 (2 hours, completed 1 month after test visit 2). Participants will be asked to collect saliva samples, to measure cortisol, immediately after they wake up on the 3 testing days. Note that testing sessions involve pupillometry (measurement of area of pupil of the eye). This is done using a specialised camera pointed at the eye and is not invasive.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 to 60 years.
* Fluent in English.
* Not currently taking any psychoactive medications (except hormone contraceptives).
* Currently meets SCID (Structured Clinical Interview for Diagnosis:DSMV) criteria for MDD--Major Depressive Disorder-- (currently depressed group only).
* Meets SCID criteria for 2 or more previous episodes of MDD, has been in remission for at least 3 months (previously depressed group only).
* No previous or current axis I diagnosis (control group only).

Exclusion Criteria:

* Previous or current diagnosis of bipolar disorder or psychotic illness.
* Previous or current anxiety disorder (control group only, anxiety disorder is permitted in current and previously depressed group as long as primary diagnosis of MDD (current or previous) is present).
* Significant suicidal ideation.
* Use of drug of abuse within the last 3 months.
* Receiving treatment (either pharmacological or psychological) for psychiatric condition.
* Medical or surgical treatment which prevents dilation/constriction of pupil.
* Prior experience of the tasks used in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptoms (self report, 16 item) | change between baseline and week 6
  Standard questionnaire measure of depressive symptoms

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms (self report, 16 item) | change between baseline and week 2
  standard questionnaire measure of depressive symptoms
Montgomery Asberg Depression Rating Scale | change from baseline to week 2 and 6
  Standard clinical rating scale for depression
Learning parameters from information bias assessment task | baseline to weeks 2 and 6
  Derived parameters from a computer based learning task (tests process presumed to be altered by IBLT-- information bias learning task-- intervention)
Salivary cortisol concentration | baseline to weeks 2 and 6
  Samples collected on waking
Learning parameters derived from pupillometry data | baseline to weeks 2 and 6
  Parameters are derived from regression of pupil size data collected during the information bias assessment task

OTHER OUTCOMES:
Speilberger State and Trait Anxiety Inventory | Baseline to weeks 2 and 6
  standard questionnaire measure of state and trait anxiety
Depressive Attributes Questionnaire | baseline to weeks 2 and 6
  Questionnaire assessing attribution bias in depression
Rumination Response Scale | baseline to weeks 2 and 6
  Questionnaire assessing tendency to ruminate
Snaith-Hamilton Pleasures Scale | Baseline to weeks 2 and 6
  Questionnaire assessing anhedonia
Accuracy and reaction time during computerised cognitive tasks | baseline to weeks 2 and 6
  Scores are derived from computer based tasks assessing emotional perception and learning

CONTACTS AND LOCATIONS:
Overall Officials: Michael Browning, MB.BS, Principal Investigator — University of Oxford
Locations (1):
- Dept of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with researchers who contact the PI after study completion.